CLINICAL TRIAL: NCT05601648
Title: SV2A Marker of Synaptogenesis in a Clinical Trial of Psilocybin for Depression
Brief Title: PET Synaptogenesis After Psilocybin In DEpression Recovery
Acronym: PET-SPIDER
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to negative results in similar trials using 11C-UCB-J
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WashU20220654925
Record Dates: First submitted 2022-10-17; First posted 2022-11-01 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Major Depressive Disorder; Anhedonia
Keywords: Psilocybin; 11C-UCB-J; SV2A
MeSH Terms: conditions — Depressive Disorder, Major; Anhedonia | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: Open label treatment study, no placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Psilocybin (Experimental): Eligible adults to undergo a single drug session with psilocybin (25mg tablet) plus supportive psychotherapy
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Psilocybin (25mg tablet) plus supportive psychotherapy

SUMMARY:
Participants with depression will be given a single dose of psilocybin and supportive psychotherapy before, during, and after drug administration. Participants will undergo positron emission tomography (PET) imaging before and one week after psilocybin using a marker of synaptic density. This design allows us to assess the relationship between neurotrophic, and antidepressant effects produced by psilocybin.

DETAILED DESCRIPTION:
The investigators are studying the neurotrophic effects of psilocybin using 11C-UCB-J, a PET marker for synaptogenesis. Psilocybin is a naturally occurring psychedelic and exerts perceptual effects via 5-HT2A receptor agonism. Psilocybin has gained a great deal of attention as a tool for psychiatric treatment, with clinical trials demonstrating symptom relief after a single dose that is immediate and persists for months. Recognizing the therapeutic potential of psilocybin, the US Food and Drug Administration granted breakthrough therapy status to the Usona Institute for Phase 2 testing of psilocybin in depression. Animal models suggest that psychedelics exert antidepressant effects by producing a rapid and powerful neurotrophic response in the brain.

The investigators will enroll patients with major depressive disorder and anhedonia. Participants will be given a single dose of psilocybin and supportive psychotherapy before, during, and after drug administration. Participants will undergo PET imaging before and one week after drug using 11C-UCB-J, a radiotracer that binds to SV2A - a marker of synaptic density and synaptogenesis. This design allows the investigators to assess the relationship between neurotrophic, and antidepressant effects produced by psilocybin.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between 18 and 65 years of age;
2. Able to provide informed consent
3. Women of childbearing age must agree to be on two forms of contraception and men are required to utilize at least one form of contraception
4. Willingness to comply and be available for all study requirements, including psychological, cognitive, and imaging for the duration of the study
5. Meeting DSM-5 criteria for major depressive disorder and current depressive episode
6. Snaith-Hamilton Anhedonia Pleasure Scale (SHAPS) ≥ 6 points
7. Willing and able to taper and/or discontinue current psychotropic medications

Exclusion Criteria:

1. Women who are pregnant or who intend to become pregnant or nurse during the study duration.
2. Presence of psychiatric conditions that are contraindications to psilocybin exposure (e.g., personal or first degree relative with history of schizophrenia spectrum or bipolar disorder);
3. Use of psychotropic medication that may interact with psilocybin (TCA, MAOi, antipsychotic/neuroleptics, anti-epileptic/mood stabilizer, lithium, SSRI, SNRI, Mirtazapine, Buproprion, Vortioxetine).
4. Recent use of psychedelics (psilocybin, LSD, ayahuasca, mescaline; past 5 years); or prior severe adverse reactions to psychedelics
5. Active suicidal ideation or history of a suicide attempt.
6. Presence of medical conditions that are contraindications to psilocybin exposure (e.g., neurological conditions or severe hypertension, severe and/or unstable metabolic or cardiovascular conditions);
7. Current medical conditions that are known to increase risk of severe coronavirus infection or deemed by a study physician to put an individual at high risk (i.e., cancer, COPD, obesity, immunosuppression, type 2 diabetes, serious heart conditions, sickle cell disease, asthma);
8. Presence of contraindications to PET or MRI scanning (renal disease, implantable devices, bone hardware, some IUDs);
9. Body mass index >30 (due to MRI confounds).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Synaptogenesis in hippocampus | 7 days after psilocybin
  Change in 11C-UCB-J signal in the hippocampus from baseline to post-treatment PET scans.
Synaptogenesis in medial prefrontal cortex | 7 days after psilocybin
  Change in 11C-UCB-J signal in the medial prefrontal cortex from baseline to post-treatment PET scans.

SECONDARY OUTCOMES:
Change in major depressive disorder symptoms | 7 days after psilocybin
  Change in Montgomery-Asberg Depression Rating Scale (MADRS) - score range 0-60 (higher score equals greater severity of depressive symptoms).
Change in anhedonia symptoms | 7 days after psilocybin
  Change in Snaith-Hamilton Anhedonia Pleasure Scale (SHAPS) - is a 14 item self-report measure assessing pleasure response/hedonic experience across domains. The SHAPS measures both anticipation and experience of pleasure. A score is obtained by making binary (disagree/strongly disagree =1) and summing the 14 items - range 0-14, greater than 3 is considered abnormal.

OTHER OUTCOMES:
Limbic functional connectivity, measured with resting state functional MRI | 7 days after psilocybin
  Resting state functional connectivity magnetic resonance imaging measures fluctuations in blood oxygenation level dependent (BOLD) signal in the brian. Functional connectivity (FC) analysis measures correlation in BOLD signal between brain areas.
  FC studies of depression have suggested pathological hyperconnectivity between cortical regions involved in mood and emotion (subgenual anterior cingulate, or sgACC), and the sense of self and rumination (default mode network or DMN). Identifying correlates of neurotrophic stimulation with rsfMRI would be of tremendous value. By acquiring concurrent PET + MRI in the same subjects the investigators will directly test the viability limbic FC as a surrogate marker of synaptogenesis (measured by PET).

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided